CLINICAL TRIAL: NCT06343090
Title: Pragmatic Clinical Trial of CD19 and CD22 CAR T-cell Sequential Therapy Versus Single CD19 CAR T-cell Bridging to Transplantation for Patients With Refractory or Relapsed B-cell Acute Lymphoblastic Leukemia
Brief Title: Clinical Trial of CD19 and CD22 CAR Sequential Therapy Versus Single CD19 CAR Bridging to HSCT for r/r B-ALL Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: The General Hospital of Western Theater Command (Other); Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai (Other); Shanghai Liquan Hospital (Other); Ruijin Hospital (Other); Central People's Hospital of Zhanjiang (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2023-003
Record Dates: First submitted 2024-03-08; First posted 2024-04-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-02

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia, in Relapse; Refractory Acute Lymphoid Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: a prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-1: CD19 CAR T and CD22 CAR T-cell sequential treatments (Sequential CAR) (Experimental)
  Interventions: Drug: CD19 CAR T-cell; Drug: CD22 CAR T cells
- Arm-2: CD19 CAR T-cell treatment bridging to HSCT (CAR+HSCT) (Experimental)
  Interventions: Drug: CD19 CAR T-cell; Procedure: hematopoietic stem-cell transplantation

INTERVENTIONS:
Drug: CD19 CAR T-cell — Murine-derived CD19 CAR T cells
Drug: CD22 CAR T cells — humanized CD22 CAR T cells
  Arms: Arm-1: CD19 CAR T and CD22 CAR T-cell sequential treatments (Sequential CAR)
Procedure: hematopoietic stem-cell transplantation — allo-HSCT
  Arms: Arm-2: CD19 CAR T-cell treatment bridging to HSCT (CAR+HSCT)

SUMMARY:
This is a multi-center, open-label, non-randomized, two-arm, non-inferior trial. Patients with r/r B-ALL would be assigned to the CD19 CAR and CD22 CAR T-cell sequential infusion group (Sequential CAR, Arm-1) and the CD19 CAR T-cell infusion bridging to hematopoietic stem cell transplantation group (CAR+HSCT, Arm-2), according their own discretion. Patients would be also allowed to assigned to the CD19 CAR T-cell infusion without consolidation therapies group (Single CAR, additional placebo arm) according their own discretion. The primary objective is to prospectively evaluate and compare the efficacy of CD19 CAR and CD22 CAR T cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT in the treatment of r/r B-ALL. The primary endpoint is event-free survival of children and adolescent and young adult (AYA) with r/r B-ALL a treated with CD19 CAR and CD22 CAR T-cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT. A total number of 353 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who meet all the following criteria can be included in the group:

  1. Patients who were diagnosed as primary refractory or relapsed B-ALL. (Criterion-reference: NCCN, version 2.2023); All the patients matched the diagnostic criteria of ALL according to the NCCN guideline (≥20% bone marrow lymphoblasts on hematopathology review of bone marrow aspirate and biopsy materials, which were confirmed by comprehensive flow cytometric immunophenotyping, minimal residual disease analysis and karyotyping of G-banded metaphase chromosomes). Molecular characterization could be obtained via interphase fluorescence in situ hybridization (FISH) testing, reverse transcriptase polymerase chain reaction (RT-PCR) testing, comprehensive testing by next-generation sequencing (NGS) for gene fusions and pathogenic mutations, etc. Determination of the World Health Organization ALL subtypes and cytogenetic and clinical risk groups were also allowed. B-ALL patients who did not achieve a complete remission after previous therapy (including the various treatment response scenarios shown in Table 1), who did not achieve a complete remission after at least two lines of TKI agents (including the various treatment response scenarios shown in Table 1), or who had ≥1 relapses were defined as having refractory or relapsed disease. Patients who were diagnosed as CD19- and CD22-positive high-risk B-ALL with continuous positive minimal residual disease (MRD) for more than three months after last therapy were also eligible. Patients had positive CD19 and CD22 expression on leukemia blasts by FCM (>80% CD19 and CD22 positive);
  2. Age from 1 to 70 years old;
  3. No serious allergic constitution;
  4. Eastern Cooperative Oncology Group (ECOG) performance status (Oken et al., 1982) score 0 to 2;
  5. Have life expectancy of at least 60 days based on investigator's judgement;
  6. Voluntary informed consent is signed by self-aware patients aged 8-70 years and by legal representatives (guardians) of pediatric patients under 18 years of age.

Exclusion Criteria:

* Patients with at least one of the following conditions are excluded:

  1. Intracranial hypertension or unconscious;
  2. Acute heart failure or severe arrhythmia;
  3. Acute respiratory failure;
  4. Other types of malignant tumors;
  5. Diffuse intravascular coagulation;
  6. Serum creatinine and/or blood urea nitrogen over 1.5 times the normal value;
  7. Sepsis or other uncontrolled infection;
  8. Uncontrolled diabetes mellitus;
  9. Severe psychological disorder;
  10. Obvious cranial lesions by cranial MRI;
  11. More than 20 leukemic cells/μL in cerebrospinal fluid;
  12. More than 30% leukemic cells in the peripheral blood;
  13. Organ recipients;
  14. Pregnant or breastfeeding;
  15. Active, uncontrolled infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or treponema pallidum (TP).

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 353 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2042-12-01 (Estimated); Study Completion 2043-09-30 (Estimated)

PRIMARY OUTCOMES:
EFS in CD19 CAR and CD22 CAR-T sequential infusion (Sequential CAR group) and CD19 CAR T-cell infusion bridging to HSCT (CAR+HSCT group) | 2-year EFS rate
  Event-free survival (EFS) of children and adolescent and young adult (AYA) with r/r B-ALL treated with CD19 CAR and CD22 CAR T-cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT.
  EFS is defined as the time from CD19 CAR T-cell infusion to the earliest relapse, death from any cause, or treatment failure.

SECONDARY OUTCOMES:
ORR in Sequential CAR group and CAR+HSCT group | 3 months (± 1 week) ORR
  Overall response rate (ORR) includes minimal residual disease-negative CR, CRh, CRi, MLFS, aplastic marrow for blood and bone marrow; central nervous system (CNS) remission; CR for lymphomatous extramedullary disease at 3 months (± 1 week) post CD19 CAR T-cell infusion in patients treated by CD19 CAR and CD22 CAR T cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT.
DOR in Sequential CAR group and CAR+HSCT group | from enrollment to the end of treatment at 15 years
  Duration of remission (DOR) of children and AYA with r/r B-ALL treated by CD19 CAR and CD22 CAR T cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT.
  DOR is defined as the time interval from the earliest qualifying minimal residual disease-negative response [i.e. CR, CRh, CRi, MLFS, or aplastic marrow (patients with blood and bone marrow disease), CNS remission (patients with CNS disease) and complete resolution of the lymphomatous enlargement by CT or PET-CT negative (for patients with a previous positive PET-CT) (patients with lymphomatous extramedullary disease)] to the date of relapse or death from any cause.
OS in Sequential CAR group and CAR+HSCT group | from enrollment to the end of treatment at 15 years
  Overall survival (OS) of children and AYA with r/r B-ALL treated by CD19 CAR and CD22 CAR T cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT.
  OS is defined as the time from CD19 CAR T-cell infusion to death from any cause.
Adverse events (AEs) in Sequential CAR group and CAR+HSCT group | from enrollment to the end of treatment at 2 years
  Total number, incidence and severity of adverse events (AEs) in patients of CD19 CAR and CD22 CAR T-cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT in the treatment of r/r B-ALL. The AEs will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus.
Levels of CD19 and CD22 CAR-T cells in Sequential CAR group | from CD19 CAR T-cell infusion to the end of treatment at 15 years
  The levels of CD19 and CD22 CAR-T cells in peripheral blood from patients treated by CD19 CAR and CD22 CAR T cell sequential infusions will be measured by flow cytometry.
Levels of CD19 CAR-T cells in CAR+HSCT group | from CD19 CAR T-cell infusion to the end of treatment at 15 years
  The levels of CD19 CAR-T cells in peripheral blood from patients in CAR+HSCT group will be measured by flow cytometry.
Levels of CD19 and CD22 CAR transgene in Sequential CAR group | from CD19 CAR T-cell infusion to the end of treatment at 15 years
  The levels of CD19 and CD22 CAR transgene in peripheral blood from patients treated by CD19 CAR and CD22 CAR T cell sequential infusions will be measured by quantitative polymerase chain reaction (qPCR).
Levels of CD19 CAR transgene in CAR+HSCT group | from CD19 CAR T-cell infusion to the end of treatment at 15 years
  The levels of CD19 CAR transgene in peripheral blood from patients in CAR+HSCT group will be measured by quantitative polymerase chain reaction (qPCR).
Quantification of B cells in Sequential CAR group and CAR+HSCT group | from enrollment to the end of treatment at 15 years
  Quantification of B cells in peripheral blood from patients treated by CD19 CAR and CD22 CAR T cell sequential infusions and CD19 CAR T-cell infusion bridging to HSCT will be measured by complete blood count and flow cytometry.

OTHER OUTCOMES:
EFS in CD19 CAR T-cell infusion without consolidation therapies (Single CAR group) | 2-year EFS rate
  EFS of children and adolescent and young adult (AYA) with r/r B-ALL treated with CD19 CAR T-cell infusion without consolidation therapies.
DOR in Single CAR group | from enrollment to the end of treatment at 15 years
  DOR of children and adolescent and young adult (AYA) with r/r B-ALL treated with CD19 CAR T-cell infusion without consolidation therapies.
OS in Single CAR group | from enrollment to the end of treatment at 15 years
  OS of children and adolescent and young adult (AYA) with r/r B-ALL treated with CD19 CAR T-cell infusion without consolidation therapies.
ORR in Single CAR group | 3 months (± 1 week) ORR
  ORR at 3 months (± 1 week) post CD19 CAR T-cell infusion, of children and adolescent and young adult (AYA) with r/r B-ALL treated with CD19 CAR T-cell infusion without consolidation therapies.
Adverse events (AEs) in Single CAR group | from enrollment to the end of treatment at 2 years
  Total number, incidence and severity of adverse events (AEs) in patients treated by CD19 CAR T-cell infusion without consolidation therapies in the treatment of r/r B-ALL. The AEs will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus.
Levels of CD19 CAR-T cells in Single CAR group | from CD19 CAR T-cell infusion to the end of treatment at 15 years
  The levels of CD19 CAR-T cells in peripheral blood from patients treated by CD19 CAR T-cell infusion without consolidation therapies will be measured by flow cytometry.
Levels of CD19 CAR transgene in Single CAR group | from CD19 CAR T-cell infusion to the end of treatment at 15 years
  The levels of CD19 CAR transgene in peripheral blood from patients treated by CD19 CAR T-cell infusion without consolidation therapies will be measured by quantitative polymerase chain reaction (qPCR).
Quantification of B cells in Single CAR group | from enrollment to the end of treatment at 15 years
  Quantification of B cells in peripheral blood from patients treated by CD19 CAR T-cell infusion without consolidation therapies will be measured by complete blood count and flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No